CLINICAL TRIAL: NCT00015041
Title: PK 0396 - Buprenorphine Dose Escalation Trial
Brief Title: Buprenorphine Dose Escalation Trial for Treatment of Non-Dependent Opiate Users - 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Cincinnati MDRU (Other)
Purpose: Treatment
Other Study IDs: NIDA-5-0012-2; Y01-5-0012-2
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1998-07

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate the effect, pharmacokinetics and dose proportionality of buprenorphine when administered to non-dependent opiate users. 1) To evaluate whether plasma concentrations of buprenorphine increase proportionally to buprenorphine dose. 2) To evaluate the dose-response of subjective and physiological effects of buprenorphine; and 3) To determine the safety of buprenorphine.

DETAILED DESCRIPTION:
This will be an open-label, single dose-escalation trial. A total of 24 opiate experienced, but not dependent subjects will receive four ascending doses of buprenorphine, 4, 8, 16, and 24 mg, respectively, with an at least a 14 day washout interval between treatments. The four treatments are sublingual administration of:

1. two 2-mg buprenorphine sublingual tablets,
2. one 8-mg buprenorphine sublingual tablet,
3. two 8-mg buprenorphine sublingual tablets; and
4. three 8-mg buprenorphine sublingual tablets.

The dose proportionality in plasma profiles of buprenorphine and dose response of the buprenorphine sublingual tablets are evaluated at buprenorphine dose range of 4 to 24 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female of any race, between 21 and 45 years of age.
2. Weigh within 15% of ideal body weight for height according to the current life insurance table.
3. Be in good physical and mental health as judged by interview and physical examination.
4. Have no significant oral cavity pathology including excessive caries, gingivitis, infectious or inflammatory disease, or recent piercing of the oral cavity.
5. Be experienced in illicit use of opiates but not be physically dependent on opiates and other drugs (except nicotine or caffeine) at the time of the study. A history of other psychoactive drug use is acceptable but preference will be for subjects reporting less frequent and more controlled illicit drug use.
6. For female subjects, test nonpregnant and use adequate birth control, and not be lactating.
7. Be capable of providing written informed consent to participate in this study.
8. Be able to comply with protocol requirements and be likely to complete all four study treatments.

Exclusion Criteria:

1. Have a diagnosis of drug addiction (other than nicotine, caffeine, and opiate) as per DSM-IV criteria.
2. Have any significant, active medical or psychiatric illnesses (other than drug dependence) which might inhibit their ability to complete the study or might be complicated by administration of study medications.
3. Have clinically significant abnormal laboratory measurements in liver function tests (AST and ALT levels greater than 3 times the upper limit of normal), hematology (CBC, differential, platelet count), serum chemistries (SMA-24) and urinalysis at screening.
4. Test positive on the HIV blood screen.
5. Have a history of significant hepatic, renal, endocrine, cardiac, nervous, psychiatric, gastrointestinal, pulmonary, hematologic or metabolic disorders.
6. Have known hypersensitivity to buprenorphine and its derivatives or opiates or opiate-like analgesics.
7. Receive any medications for medical conditions.
8. Have any condition or history considered by the investigator(s) to place the subjects at increased risk.
9. Do not actively meet the inclusion criteria at the time of screening.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-11; Primary Completion 1998-06 (Actual); Study Completion 1998-07 (Actual)

PRIMARY OUTCOMES:
PK parameters of buprenorphine
Intoxication and withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Somoza, M.D., Ph.D., Principal Investigator — Cincinnati MDRU
Locations (1):
- Cincinnati MDRU, Cincinnati, Ohio, United States